CLINICAL TRIAL: NCT01605669
Title: Correlation of Auscultatory Severity of Aortic Stenosis With Trans Thoracic Echocardiography
Acronym: Cassette
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: 3M (Industry); The Geneva Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2011.0123
Record Dates: First submitted 2012-05-17; First posted 2012-05-25 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Stenosis
Keywords: Auscultation; Aortic stenosis; computer assisted auscultation; Aortic Stenosis Acceleration Index
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic stenosis patients: Patients with varying degrees of aortic stenosis without significant additional valvular disease will be considered eligible for this study. All participants will recieve a transthoracic echocardiogram and recorded cardiac auscultation.
  Interventions: Other: Tranthoracic Echocardiogram; Device: Cardiac Ascultation Recordings with Electronic stethoscope

INTERVENTIONS:
Other: Tranthoracic Echocardiogram — standard measurement
Device: Cardiac Ascultation Recordings with Electronic stethoscope — 3M device

SUMMARY:
According to the 2006 ACC/AHA practice guidelines for valvular heart disease, patients with asymptomatic aortic stenosis(AS) should have screening transthoracic echocardiograms (TTE) performed annually for severe disease, every 1-2 years for moderate disease and every 3-5 years for mild disease. This results in a multitude of screening studies in the investigators patient population. 3M has developed a new stethoscope and phonocardiography software capable of identifying the peak intensity of the AS murmur and tracking it as it moves towards the second heart sound potentially indicating increasing severity of disease. Currently there exists no data to demonstrate that the aortic stenosis acceleration index (ASAI) correlates to disease severity or progression of disease. The ASAI measures the timing of the peak intensity of the systolic murmur and compares it to the total time in systole (S2-x/s2-s1) where s1 is the first heart sound; S2 is the second heart sound and x with the time between S1 and the peak intensity of the murmur. In this study the investigators propose to correlate the ASAI to standard TTE measurements of aortic stenosis severity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years of age and older.
2. Subjects must have asymptomatic Aortic Stenosis documented by prior echocardiographic examination.
3. Subjects must be able to sit for auscultation examination.
4. Subject must be able to complete a TTE .
5. Subjects must voluntarily agree to participate in the study and sign the informed consent and healthcare information authorization forms.

Exclusion Criteria:

1. Subjects with significant additional valvular heart disease.
2. Subjects with unrecordable heart sounds.
3. Subjects with known or who may have been previously diagnosed with congenital heart disease.
4. Subjects with atrial fibrillation.
5. Subjects with history of cardiac surgery.
6. Subjects who have conditions which the researcher feels may limit the recordability of the heart sounds or the accuracy of the echocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Aortic Stenosis seen in the internal medicine clinic at NMCSD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Bennett, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BRAUNWALD E, GOLDBLATT A, AYGEN MM, ROCKOFF SD, MORROW AG. Congenital aortic stenosis. I. Clinical and hemodynamic findings in 100 patients. II. Surgical treatment and the results of operation. Circulation. 1963 Mar;27:426-62. doi: 10.1161/01.cir.27.3.426. No abstract available. PMID 14015087
- [Background] Bonner AJ Jr, Sacks HN, Tavel ME. Assessing the severity of aortic stenosis by phonocardiography and external carotid pulse recordings. Circulation. 1973 Aug;48(2):247-52. doi: 10.1161/01.cir.48.2.247. No abstract available. PMID 4726205
- [Background] Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; 2006 Writing Committee Members; American College of Cardiology/American Heart Association Task Force. 2008 Focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1998 Guidelines for the Management of Patients With Valvular Heart Disease): endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Circulation. 2008 Oct 7;118(15):e523-661. doi: 10.1161/CIRCULATIONAHA.108.190748. Epub 2008 Sep 26. No abstract available. PMID 18820172
- [Background] Stewart BF, Siscovick D, Lind BK, Gardin JM, Gottdiener JS, Smith VE, Kitzman DW, Otto CM. Clinical factors associated with calcific aortic valve disease. Cardiovascular Health Study. J Am Coll Cardiol. 1997 Mar 1;29(3):630-4. doi: 10.1016/s0735-1097(96)00563-3. PMID 9060903

RESULTS

PARTICIPANT FLOW:
Groups:
- Aortic Stenosis Patients: Patients with varying degrees of aortic stenosis without significant additional valvular disease will be considered eligible for this study.
Period: Overall Study
Arm/Group | Aortic Stenosis Patients
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aortic Stenosis Patients
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Aortic Stenosis Acceleration Index Compared to Aortic Stenosis Severity
Description: The ASAI measures the timing of the peak intensity of the systolic murmur and compares it to the total time in systole (S2-x/s2-s1) where s1 is the first heart sound; S2 is the second heart sound and x with the time between S1 and the peak intensity of the murmur. Aortic Stenosis severity will be measured by peak and mean aortic valve gradients as well as aortic valve area derived from the continuity equation. ASAI was averaged and compared to the mean aortic gradient. ROC curve was calculated for ASAI predicting a mean gradient of >30mmHg. ASAI of 34 was determined to provide the optimal combination of specificity and sensitivity and therefore set as the cut off point for significant Aortic Stenosis.
Time Frame: There is a single measurement taken on the day of enrollment. The ascultatory recording and echocardiogram will occur at the same visit. There will be no additional visits or study followup.
Measure: Number; unit: participants
Groups:
- Mean Pressure Gradient >=30mmHg (Positive): Patients with varying degrees of aortic stenosis without significant additional valvular disease will be considered eligible for this study.
Arm/Group | Mean Pressure Gradient >=30mmHg (Positive) | Mean Pressure Gradient <30mmHg (Negative)
Number analyzed (Participants) | 22 | 14
participants
  ASAI >= 34 (positive) | 21 | 8
  ASAI < 34 (negative) | 1 | 6
Statistical Analysis 1: Comparison: Mean Pressure Gradient >=30mmHg (Positive); Test type: Superiority or Other; Percentage Sensitivity = 85.7
Statistical Analysis 2: Comparison: Mean Pressure Gradient <30mmHg (Negative); Test type: Superiority or Other; Percent Specificity = 72.4
Statistical Analysis 3: Comparison: Mean Pressure Gradient >=30mmHg (Positive) vs Mean Pressure Gradient <30mmHg (Negative); Test type: Superiority or Other; Percent Error Rate = 25 — Error rate of 9/36 is equal to total of false positives plus false negatives over the total of participants analyzed

ADVERSE EVENTS:
Arm/Group | Aortic Stenosis Patients
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
Patients with significant concomitant valvular disease were not evaluated. The software does not provide immediate feedback on the severity of the stenosis. Multiple early recordings had artifact noise rquiring modificaiton of recording techniques.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No